CLINICAL TRIAL: NCT06254742
Title: Study on Preference and Safety of HHPG-19K Injection and Auto-HHPG-19K Injection in Prevention of Chemotherapy-related Moderate to Severe Neutropenia of Patients With Nonmyeloid Malignancies
Brief Title: A Trial of HHPG-19K Injection and Auto-HHPG-19K Injection in Prevention of Chemotherapy-related Moderate to Severe Neutropenia of Patients With Nonmyeloid Malignancies
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor's R&D strategy is adjusted.
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Auto-HHPG-19K-301
Record Dates: First submitted 2024-01-21; First posted 2024-02-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Patients With Nonmyeloid Malignancies Receiving Antineoplastic Therapy Based on Chemotherapy Regimens at Moderate to High Febrile Neutropenia (FN) Risk
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): first cycle: Auto-HHPG-19K Injection second cycle: HHPG-19K Injection
  Interventions: Drug: HHPG-19K Injection
- Treatment group B (Experimental): first cycle: HHPG-19K Injection second cycle: Auto-HHPG-19K Injection
  Interventions: Drug: HHPG-19K Injection

INTERVENTIONS:
Drug: HHPG-19K Injection — first cycle: Auto-HHPG-19K Injection or HHPG-19K Injection second cycle: HHPG-19K Injection or Auto-HHPG-19K Injection

SUMMARY:
The study is being conducted to evaluate the preference, and safety of HHPG-19K Injection and Auto-HHPG-19K Injection in Prevention of chemotherapy-related moderate to severe neutropenia of Patients with nonmyeloid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. The patient signs the informed consent form and voluntarily participate in this study;
2. Age ≥18 years;
3. Have the ability to read and understand Chinese;
4. Pathologically or histologically confirmed diagnosis of non-myeloid malignant tumor diseases (including solid tumors and malignant hematologic tumors);
5. Patients who plan to receive at least two consecutive cycles of anti-tumor trerapy based on a moderate to high FN risk chemotherapy regimen (see Appendix 4 for details of the chemotherapy regimen);
6. The investigator determines that the patient are eligible to receive administration of HHPG-19K injection and Auto-HHPG-19K injection (delivered through an adhesive patch automatic drug delivery device);
7. ECOG (Eastern Cooperative Oncology Group score) score 0-1 points;
8. Expected survival ≥3 months;
9. Good function of major organs, meeting the following criteria:

   1. Neutrophil count ≥1.5 ×109/L;
   2. Platelet count≥75 ×109/L;
   3. Hemoglobin level≥80 g/L.
10. Women of childbearing age must take a blood pregnancy test within 3 days before randomization, and the result is negative, and they should not be lactating. Female subjects of childbearing age and male subjects whose partners are women of childbearing age must agree to approach highly effective contraceptive methods from the day of signing the informed consent form until at least 6 months after the last administration (for female subjects) or 3 months after the last administration (for male subjects).

Exclusion Criteria:

1. Women who are planning to become pregnant or breastfeeding;
2. Allergic to polyacrylate adhesives, HHPG-19K, polyethylene glycol recombinant human granulocyte stimulating factor, recombinant human granulocyte stimulating factor and other preparations expressed in Escherichia coli;
3. Having a history of bone marrow transplantation and/or stem cell transplantation;
4. Other situations deemed unsuitable for inclusion in the study as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The preference ratio of patients for HHPG-19K and Auto-HHPG-19K , as assessed in the Patient Preference Questionnaire"Considering your overall experience in this study, which administration method do you prefer for drug injection?" | Evaluation after administration on Day 2 of Cycle 2 (each cycle is approximately 21 days)
  The available options for a participant's response were HHPG-19K, Auto-HHPG-19K, and No preference.

SECONDARY OUTCOMES:
The preference ratio of physicians and nurses for HHPG-19K and Auto-HHPG-19K, according to the question in the "Preference Questionnaire of Physician and Nurse": "Which formulation would you recommend for patient use?" | approximately 2 months
  The available options for a participant's response were HHPG-19K, Auto-HHPG-19K, and No preference.
Factors influencing patients' preference for HHPG-19K and Auto-HHPG-19K. | Evaluation after administration on Day 2 of Cycle 2 (each cycle is approximately 21 days).
  According to participants' response in the Patient Preference Questionnaire and the Patient Satisfaction Questionnaire, conducting descriptive summaries of influencing factors, including physical condition, convenience, injection pain, and individual evaluation. The available options for a participant's response in the Patient Satisfaction Questionnaire were No, a little, quite, and extremely. The available options for a participant's response in the Patient Preference Questionnaire were HHPG-19K, Auto-HHPG-19K, and No preference.
Factors influencing the preference of physician and nurse for HHPG-19K and Auto-HHPG-19K | Evaluation after experiencing at least 3 cases of HHPG-19K injection and 3 cases of Auto-HHPG-19K injection therapy
  Influencing factors were analysed according to the items in the Preference Questionnaire of Physician and Nurse.
The injection experience of patients using HHPG-19K and Auto-HH PG-19K | Evaluation after administration on Day 2 of Cycle 2 (each cycle is approximately 21 days)
  Conduct descriptive summaries based on the patient's injection experience items in the Patient Satisfaction Questionnaire. The available options for a participant's response in the Patient Satisfaction Questionnaire were No, a little, quite, and extremely.
The proportion of successful administration of HHPG-19K Injection within 24h-72h after the end of chemotherapy drugs. | Evaluation after administration on Day 2 of Cycle 2 (each cycle is approximately 21 days)
  The proportion was summarized based on the time of HHPG-19K administration for each patient.
Incidence of adverse events Auto-HHPG-19K Injection. | From screening period to the last follow-up visit(approximately up to 2 months )
  Adverse events were assessed by CTCAE v5.0

IPD SHARING:
Plan to Share IPD: Undecided